CLINICAL TRIAL: NCT02806739
Title: A Pilot Study of Soy Protein and Isoflavone Supplementation for Improved Glucose Metabolism and Lipid Profiles in Pregnant Women at High Risk for Gestational Diabetes Mellitus (GDM)
Brief Title: Soy Supplementation and Gestational Diabetes
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Massachusetts, Boston (Other)
Collaborators: University of Massachusetts, Worcester (Other); Tufts University (Other); Hallmark Health System (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UL1TR000161 (NIH)
Record Dates: First submitted 2013-01-22; First posted 2016-06-21 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2016-10

CONDITIONS: Gestational Diabetes
Keywords: Soy protein; isoflavones; gestational diabetes
MeSH Terms: conditions — Diabetes, Gestational | interventions — Soybean Proteins; Isoflavones; Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Soy Group (Soy Protein + Isoflavones) (Experimental): Intervention: Soy-based whole foods containing about 25 grams of soy protein and 60-75 mg isoflavones.
  Intervention group will consume soy foods containing about 25 grams of soy protein and 60-75 mg isoflavones per day, from 16th gestational week to birth. Examples of soy foods that contain 25 grams of soy protein and 60-75mg isoflavones include: 2 cups of soy milk, or 12 ounces tofu, or a half cup of soy nuts. Women in the Soy Group will be instructed by a registered dietitian how to incorporate the soy foods into their daily diet.
  Interventions: Dietary Supplement: Soy Group (Soy Protein + Isoflavones)
- Control Group (Minimize Soy Intake) (Placebo Comparator): Control Group will avoid soy supplements and minimize intake of soy foods.
  Interventions: Dietary Supplement: Control Group (Minimize Soy Intake)

INTERVENTIONS:
Dietary Supplement: Soy Group (Soy Protein + Isoflavones) — Women in the intervention group are asked to eat a combination of soy foods that contain about 25 grams of protein and 60-75 milligrams of isoflavones per day, from the 16th gestational week to birth. A registered dietitian will instruct them to incorporate the soy foods into their daily diet.
  Arms: Soy Group (Soy Protein + Isoflavones)
Dietary Supplement: Control Group (Minimize Soy Intake) — Women in the control group will be instructed by the dietitian how to avoid soy supplements and minimize soy intake.
  Arms: Control Group (Minimize Soy Intake)

SUMMARY:
The purpose of this study is to assess the feasibility of randomizing pregnant women at high risk for gestational diabetes to a 24-week period of soy food consumption. This study will also examine the effects of soy protein and isoflavones on glucose metabolism and lipid levels among pregnant women at high risk for gestational diabetes, and on child's weight and height at birth and 6 weeks of life.

DETAILED DESCRIPTION:
Evidence from animal studies, human observational studies, and some randomized controlled trials has suggested that soy protein and isoflavones have beneficial effects on lipid and glucose metabolism. Additionally, soy isoflavones can diffuse across the placenta, enter fetal circulation and potentially reduce the susceptibility to cardiometabolic disorders in adulthood. Given the high prevalence of GDM and its serious health consequences for women and their children, and likely health benefits of soy protein and isoflavones on a panel of metabolic parameters, the role of maternal supplementation of soy protein and isoflavones for prevention of GDM and/or minimization of GDM severity in mothers and for improving health indicators in their offspring merits investigation.

This study will provide new and essential information about the efficacy and feasibility of using soy-based whole foods to prevent and manage gestational diabetes development. This study will be a randomized, placebo-controlled trial. Forty pregnant women at high risk for gestational diabetes will be recruited from the obstetrics services at the Melrose Wakefield Hospital and Tufts Medical Center, and randomized to receive soy-based foods or minimize soy intake, from the 16th gestational week to birth. To measure participants' compliance with the treatment, the study will use three methods: (1) monthly telephone interview about adherence to the treatment; (2) daily soy food intake log; and (3) serum isoflavone concentrations. To evaluate the effects of soy supplementation on GDM, the study will collect blood samples to measure glucose, insulin, HbA1c, and lipids (triglycerides, total cholesterol, high-density lipoprotein cholesterol and low-density lipoprotein cholesterol ). The study will also measure weight and body composition of participating pregnant women and the participants' respective children's weight, length and body composition.

ELIGIBILITY:
Inclusion Criteria:

* Age >=18 years
* ≤ 18 weeks of pregnancy
* Singleton pregnancy
* Have at least one of the risk factors for GDM, including overweight (BMI ≥ 25 kg/m2) before this pregnancy, first-degree relative with type-2 diabetes mellitus (T2DM), abnormal glucose tolerance/GDM in previous pregnancy, and/or history of macrosomia (birth weight ≥ 4,000 gram) in previous pregnancy
* Being able and willing to give written informed consent.

Exclusion Criteria:

* Allergic to soy or milk products
* Current smoker
* Preexisting diabetes outside of pregnancy or other heath conditions that could affect glucose levels
* Chronic or serious medical conditions such as hypertension, heart disease, stroke, chronic renal or hepatic disease, or malignant disease (by self-report and medical record review)
* Use of medications that could interfere with insulin secretion or insulin sensitivity
* Weight loss during this pregnancy more than 10% of pre-pregnancy body weight
* Current severe nausea and/or vomiting (by self-report).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-01; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Adverse Events That Are Related to Treatment | From enrollment through study completion, an average of 30 weeks or 210 days.
  The first aim of this study is to determine the safety of soy supplementation during pregnancy. This will be assessed by the number of participants who reported adverse events that are related to the study treatment.

SECONDARY OUTCOMES:
Effects of Soy Intake on Triglycerides (TG) | Baseline (14 weeks of pregnancy), 28 weeks of pregnancy, and 6 week postpartum
  The second aim of this study is to assess the effects of soy intake during pregnancy on glucose and lipid metabolism, and inflammation. Triglycerides (TG) is one of the measurements of lipid metabolism.
Effects of Soy Intake on Total Cholesterol (TC) | Baseline (14 weeks of pregnancy), 28 weeks of pregnancy, and 6 week postpartum
  The second aim of this study is to assess the effects of soy intake during pregnancy on glucose and lipid metabolism, and inflammation. Total cholesterol (TC) is a measurement of lipid metabolism.
Effects of Soy Intake on High-density Lipoprotein Cholesterol (HDL-C) | Baseline (14 weeks of pregnancy), 28 weeks of pregnancy, and 6 week postpartum
  The second aim of this study is to assess the effects of soy intake during pregnancy on glucose and lipid metabolism, and inflammation. High-density lipoprotein cholesterol (HDL-C) is a measurement of lipid metabolism.
Effects of Soy Intake on Free Fatty Acid (FFA) | Baseline (14 weeks of pregnancy), 28 weeks of pregnancy, and 6 week postpartum
  The second aim of this study is to assess the effects of soy intake during pregnancy on glucose and lipid metabolism, and inflammation. Free fatty acid (FFA) is a measurement of lipid metabolism.
Effects of Soy Intake on Fasting Glucose | Baseline (14 weeks of pregnancy), 28 weeks of pregnancy, and 6 week postpartum
  The second aim of this study is to assess the effects of soy intake during pregnancy on glucose and lipid metabolism, and inflammation. Fasting glucose is a measurement of glucose metabolism.
Effects of Soy Intake on Fasting Insulin | Baseline (14 weeks of pregnancy), 28 weeks of pregnancy, and 6 week postpartum
  The second aim of this study is to assess the effects of soy intake during pregnancy on glucose and lipid metabolism, and inflammation. Fasting insulin is a measurement of glucose metabolism.
Effects of Soy Intake on Hemoglobin A1c (HbA1c) | Baseline (14 weeks of pregnancy), 28 weeks of pregnancy, and 6 week postpartum
  The second aim of this study is to assess the effects of soy intake during pregnancy on glucose and lipid metabolism, and inflammation. Hemoglobin A1c (HbA1c) is a measurement of glucose metabolism.
Effects of Soy Intake on C-reactive Protein (CRP) | Baseline (14 weeks of pregnancy), 28 weeks of pregnancy, and 6 week postpartum
  The second aim of this study is to assess the effects of soy intake during pregnancy on glucose and lipid metabolism, and inflammation. C-reactive protein (CRP) is a measurement of inflammation.

CONTACTS AND LOCATIONS:
Overall Officials: Ling Shi, PhD, Principal Investigator — University of Massachusetts, Boston
Locations (1):
- Tufts Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) will be not shared. Data will be shared in aggregated way in publications and national conferences.